CLINICAL TRIAL: NCT00590525
Title: Inflammation as a Predictor in Cardioversion of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Susan Schima, MD, Creighton University
Other Study IDs: 04-13547; 04-13547
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Atrial Fibrillation
Keywords: hsCRP
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Cardioversion

INTERVENTIONS:
Procedure: Cardioversion — Baseline hsCRP will be drawn the morning of, prior to, cardioversion. An EKG to document the patient's rhythm will be obtained at the one-month mark

SUMMARY:
The laboratory test, C-Reactive Protein (CRP), has become well established as a marker of inflammation. Recently a high CRP level (indicating an increase in inflammation) was identified as a risk factor for atrial fibrillation. We are conducting this study with patients such as yourself with atrial fibrillation who are planning to undergo cardioversion to determine what sort of relationship exists between CRP levels and atrial fibrillation. We will then look at success rates of converting atrial fibrillation to normal sinus rhythm, compared to patients' CRP levels.

ELIGIBILITY:
Inclusion Criteria

* Atrial fibrillation patients referred for DC cardioversion
* On stable medical therapy

Exclusion Criteria

* Known chronic inflammatory states such as infections, rheumatoid arthritis or known vasculitides.
* Patients having undergone recent surgery or who are on steroid therapy for any reason will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing DC cardioversion at The Cardiac Center electrophysiology lab who meet these criteria will be enrolled.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2004-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
We hypothesize that a higher hsCRP is associated with higher failure rates in patients undergoing cardioversion for atrial fibrillation | 1 month

SECONDARY OUTCOMES:
secondary endpoint will be if a new inflammatory disease state is diagnosed at the one-month mark. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schima, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States